CLINICAL TRIAL: NCT00833716
Title: An Open-label Trial Investigating the Pharmacokinetics and the Tolerability of NN9535 in Subjects With Normal Renal Function and Various Degrees of Impaired Renal Function
Brief Title: Effect of Renal Impairment on the Pharmacokinetics of NN9535
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NN9535-3616
Record Dates: First submitted 2009-01-29; First posted 2009-02-02 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2; Renal Impairment
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2; Renal Insufficiency | interventions — semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: semaglutide

INTERVENTIONS:
Drug: semaglutide — 10 mg/mL of semaglutide solution for s.c. injection, single dose
  Other Names: NN9535

SUMMARY:
This trial is conducted in the United States of America (USA). The aim of this clinical trial is to investigate how different degrees of renal impairment (mild, moderate, severe and end-stage renal disease) affect the pharmacokinetics of NN9535.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities. (Trial-related activities are any procedure that would not have been performed during normal management of the subject)
* Subjects meeting the pre-defined GFR (glomerular filtration rate) criteria (estimated by the Cockcroft & Gault formula) for any of the renal function groups
* Body Mass Index (BMI) equal to or less than 40kg/m2

Exclusion Criteria:

* Known or suspected allergy to trial product(s) or related products
* Renal transplanted patients
* Certain cardiac problems (heart failure, unstable angina, MI (myocardial infarction) within the last 3 months)
* Known current hepatic dysfunction or severe hepatic disease during the last 12 months
* Female of childbearing potential/breast feeding
* History of alcoholism or drug abuse
* Blood donation during the last 8 weeks prior to the study
* Past or current history of pancreatitis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2009-02-02 (Actual); Primary Completion 2010-07-26 (Actual); Study Completion 2010-07-26 (Actual)

PRIMARY OUTCOMES:
AUC of NN9535 | at 21 days

SECONDARY OUTCOMES:
Laboratory safety, adverse events | at 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (3):
- United States (3):
  - Novo Nordisk Investigational Site, Miami, Florida
  - Novo Nordisk Investigational Site, Orlando, Florida
  - Novo Nordisk Investigational Site, Knoxville, Tennessee

REFERENCES:
- [Result] Marbury T, Flint A, Segel S, Lindegaard M, Lasseter K. Pharmacokinetics and tolerability of semaglutide, a once-weekly human GLP-1 analog, in subjects with and without renal impairment. Diabetes 2014; 63 (Suppl 1): A260 (abstract 1010-P)
- [Result] Marbury TC, Flint A, Jacobsen JB, Derving Karsbol J, Lasseter K. Pharmacokinetics and Tolerability of a Single Dose of Semaglutide, a Human Glucagon-Like Peptide-1 Analog, in Subjects With and Without Renal Impairment. Clin Pharmacokinet. 2017 Nov;56(11):1381-1390. doi: 10.1007/s40262-017-0528-2. PMID 28349386
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com